CLINICAL TRIAL: NCT03061695
Title: The Application of the Spectral Analysis and Characteristic Parameters of Digitized Respiratory Sounds in the Confirmation of the Position of the Balloon of Endobronchial Blockers - an Observational Study
Brief Title: Application of Digitized Respiratory Sounds for Confirmation of the Position of the Balloon of Endobronchial Blockers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201611044RINA
Record Dates: First submitted 2017-02-01; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Respiratory Sounds
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observation study is to evaluate the application of the spectral analysis and characteristic parameters of digitized respiratory sounds in the confirmation of the position of the balloon of endobronchial blockers

DETAILED DESCRIPTION:
This is an observational study. We will recruit 30 patients who are scheduled for thoracic surgery under general anesthesia with tracheal intubation and need endobronchial blocker for unilateral lung ventilation during the operation. The standard procedures for confirming the position of the balloon of the endobronchial blocker, including the stethoscopic inspection and the fiberoptic examination, will be performed as routine practice. But in our study, besides the above routine practice, a microphone will be connected to the distal end of the stethoscope (the microphone will not contact directly with the patients) during the checking procedure to record the breathing sound into a digital computer as electronic files. These breathing sound files will be analyzed in a later time with spectral transformation and the characteristics are extracted. These digital signal processing results will be compared with the results of fibroptic exmination and the stethoscopic auscultation in the correct rate of diagnosing the position of the endobronchial balloon. The aim of this study is to examine the usefulness of the spectral parameters of the digitalized breathing sound in confirming the position of the endobronchial blocker balloon.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic disease patients who are scheduled for thoracic surgery and lung isolation requiring endobronchial blocker placement during the surgery
* Adult patients (no younger than 20 years old)

Exclusion Criteria:

* Patients with significant thoracic diseases which result in abnormal respiratory sounds

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Thoracic patients scheduled for thoracic surgery and lung isolation during the surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-02-28 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Position of the endobronchial blocker | 1 day
  Position of the ballon of the endobronchial blocker (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Hsun Huang, MD, PhD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: Undecided